CLINICAL TRIAL: NCT07104461
Title: A Single-blind Randomised Study to Test the Effects of Protein-enriched Breakfast Meals With Varying Protein Sources Compared to a Standard Meal on the Regulation of Appetite and Satiety in Healthy Human Volunteers
Brief Title: Advanced Protein-based Program for Effective Treatment of Appetite Regulation and Obesity
Acronym: APPETITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Westminster (Other)
Responsible Party: Principal Investigator, Mohammed Gulrez Zariwala, Professor of Translational Physiology, University of Westminster
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ETH2223-1377
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Appetite and General Nutritional Disorders
Keywords: nutraceutical; protein; whey; potato protein; rice protein; pea protein; appetite; satiety; insulin; glucose; ghrelin; appetite hormone; GLP-1; PYY; GIP; supplement
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Crossover Assignment, single-blind, randomised, quadruple crossover
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Oat porridge (Sham Comparator): Control Meal (9.5 g total protein)
  Interventions: Other: Oat porridge
- Oat porridge with whey protein (Active Comparator): (total protein 40.5 g; of which whey protein isolate contributed 34.2 g of protein)
  Interventions: Dietary Supplement: Whey protein isolate
- Oat porridge with potato protein (Active Comparator): (total protein 40.6 g; of which potato protein isolate contributed 34.39 g of protein)
  Interventions: Dietary Supplement: Potato protein isolate
- Meal replacement shake (Active Comparator): (total protein 40 g, mostly from pea protein and brown rice protein isolates)
  Interventions: Dietary Supplement: Meal replacement shake

INTERVENTIONS:
Other: Oat porridge — Oat flakes, 81g (equivalent to 9 g of protein), were presented to participants in the form of porridge, prepared with 500 mL coconut milk (equivalent to 0.5 g of protein) and 10 g of zero calorie sugar free syrup.
  The total energy content was equivalent to 400 Kcal.
  Participants were instructed to consume the entire meal presented to them in 15 minutes on an empty stomach when attending the study.
  Arms: Oat porridge
Dietary Supplement: Whey protein isolate — Whey protein isolate, 38g (equivalent to 34.2 g of protein), was presented to participants in the form of a porridge.
  Other ingredients in the whey protein enriched porridge:
  * Oat flakes 54 g (equivalent to 6 g of protein)
  * Coconut milk 300 mL (equivalent to 0.3 g of protein)
  * Water 150 mL
  * Zero calorie sugar free syrup 10 g
  The total energy content was equivalent to 401.74 Kcal.
  Participants were instructed to consume the entire meal presented to them in 15 minutes on an empty stomach when attending the study
  Arms: Oat porridge with whey protein
Dietary Supplement: Potato protein isolate — Potato protein isolate, 38g (equivalent to 34.39 g of protein), was presented to participants in the form of a porridge.
  Other ingredients in the potato protein enriched porridge:
  * Oat flakes 54 g (equivalent to 6 g of protein)
  * Coconut milk 300 mL (equivalent to 0.3 g of protein)
  * Water 150 mL
  * Zero calorie sugar free syrup 10 g
  The total energy content equiv. 401.36 Kcal.
  Participants were instructed to consume the entire meal presented to them in 15 minutes on an empty stomach when attending the study.
  Arms: Oat porridge with potato protein
Dietary Supplement: Meal replacement shake — A meal replacement, 90 g (equivalent to 40 g of total protein), was presented to participants in the form of a shake.
  Other ingredients in the meal replacement shake:
  - Water 500 mL
  The total energy was equivalent to 400 Kcal
  Participants were instructed to consume the entire meal replacement shake presented to them in 15 minutes on an empty stomach when attending the study.
  Arms: Meal replacement shake

SUMMARY:
INTRODUCTION: Obesity is a global epidemic, with over 2.5 billion adults being classified as overweight and 890 million of these classified as obese. Overweight and obesity are the 5th cause of mortality globally, with an estimated 2.8 million related deaths among adults. The rising prevalence of obesity in adults is leading to a rise in the prevalence of type 2 diabetes, with an estimated 462 million individuals affected globally. At present, the most effective non-surgical obesity treatments offered by the National Health Service (NHS) are the subcutaneously administered GLP-1 receptor agonists. However, they may present potentially serious side effects following short-term use, and there are still uncertainties around long-term use side effects. Therefore, a dietary approach to weight loss or maintenance seems preferable.

Increasing protein intake is a commonly applied nutritional approach to appetite regulation. The increase in protein intake is often achieved by supplementation, using proteins isolated from dairy, such as whey and casein. However, with more individuals following plant-based diets over recent years, the interest in plant-based protein supplements has increased. While dairy-based proteins are well-characterised, the appetite regulatory characteristics of plant-based proteins have not yet been fully elucidated.

The main aim of this study is to investigate the effects of protein-enriched food items on appetite regulation compared to a standard carbohydrate-rich meal. Furthermore, this study will investigate whether there are any differences in appetite-related hormonal responses to a plant protein-containing meal replacement shake (containing rice and pea protein) or a potato protein-enriched standard carbohydrate-based meal compared to a whey protein-enriched standard carbohydrate-based meal.

DETAILED DESCRIPTION:
Intervention study with four treatment groups in a randomised, single-blind, quadruple crossover design.

Healthy male participants (between the ages of 18 to 50 years) will receive four different isocaloric intervention meals with the same mass, on separate visit days, following a minimum of 8 hours overnight fast. The four meals will contain oat porridge prepared with coconut milk as a control, oat porridge prepared with coconut milk with added whey or potato protein isolates, and a complete meal replacement shake containing plant-based pea and rice proteins. The intervention meals will be followed by a standardised pasta-based ready meal after the 3-hour observation period. All participants will observe at least a two-day washout period between the differing treatments.

Biological samples (blood) will be collected at various times during the visit. Blood samples will be collected at baseline 0 min prior (T0), then at 30 min (T30), 60 min (T60), 120 min (T120) and 180 min (T180) after the intervention meal consumption.

In addition, pertinent questionnaires, Visual Analogue Scale [VAS] for assessing satiety and VAS for assessing intervention meals' perception and palatability will be collected. VAS for the assessment of satiety will be collected at T0, T30, T60, T120 and T180 and VAS assessing the perception and palatability of the intervention meals will be collected immediately following meal consumption.

ELIGIBILITY:
Inclusion Criteria:

* Males (18-50 years of age)
* Lean and Overweight subjects (BMI 18.5 - 30 kg/m2)
* Sedentary and physically active subjects
* Healthy subjects

Exclusion Criteria:

* Female
* <18, >50 years
* Dieting
* Consumption of >14 units of alcohol/week
* Allergies to test foods/drinks
* Illnesses or on medication (with a possible effect on taste and/or appetite)
* Devices such as pacemakers
* Smokers
* Gastrointestinal disorders
* Eating disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate and meal replacement shake on glucose levels (T30) | Glucose measured 30 minutes post meal consumption
  Glucose (mmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on glucose levels (T60) | Glucose measured 60 minutes post meal consumption
  Glucose (mmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on glucose levels (T120) | Glucose measured 120 minutes post meal consumption
  Glucose (mmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on glucose levels (T180) | Glucose measured 180 minutes post meal consumption
  Glucose (mmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on insulin levels (T30) | Insulin measured 30 minutes post meal consumption
  Insulin (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on insulin levels (T60) | Insulin measured 160 minutes post meal consumption
  Insulin (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on insulin levels (T120) | Insulin measured 120 minutes post meal consumption
  Insulin (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on insulin levels (T180) | Insulin measured 180 minutes post meal consumption
  Insulin (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on glucagon-like peptide 1 levels (T30) | Glucagon-like peptide 1 measured 30 minutes post meal consumption
  Glucagon-like peptide 1 (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on glucagon-like peptide 1 levels (T60) | Glucagon-like peptide 1 measured 60 minutes post meal consumption
  Glucagon-like peptide 1 (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on glucagon-like peptide 1 levels (T120) | Glucagon-like peptide 1 measured 120 minutes post meal consumption
  Glucagon-like peptide 1 (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on glucagon-like peptide 1 levels (T180) | Glucagon-like peptide 1 measured 180 minutes post meal consumption
  Glucagon-like peptide 1 (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on gastric inhibitory polypeptide (T30) | Gastric inhibitory polypeptide measured 30 minutes post meal consumption
  Glucagon-like peptide 1 (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on gastric inhibitory polypeptide (T60) | Gastric inhibitory polypeptide measured 60 minutes post meal consumption
  Glucagon-like peptide 1 (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on gastric inhibitory polypeptide (T120) | Gastric inhibitory polypeptide measured 120 minutes post meal consumption
  Glucagon-like peptide 1 (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on gastric inhibitory polypeptide (T180) | Gastric inhibitory polypeptide measured 180 minutes post meal consumption
  Glucagon-like peptide 1 (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on peptide tyrosine tyrosine levels (T30) | Peptide tyrosine tyrosine measured 30 minutes post meal consumption
  Peptide tyrosine tyrosine (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on peptide tyrosine tyrosine levels (T60) Markers: peptide tyrosine tyrosine (pmol/L) | Peptide tyrosine tyrosine measured 60 minutes post meal consumption
  Peptide tyrosine tyrosine (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on peptide tyrosine tyrosine levels (T120) | Peptide tyrosine tyrosine measured 120 minutes post meal consumption
  Peptide tyrosine tyrosine (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on peptide tyrosine tyrosine levels (T180) | Peptide tyrosine tyrosine measured 180 minutes post meal consumption
  Peptide tyrosine tyrosine (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on ghrelin levels (T30) | Ghrelin measured 30 minutes post meal consumption
  Ghrelin (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on ghrelin levels (T60) | Ghrelin measured 60 minutes post meal consumption
  Ghrelin (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on ghrelin levels (T120) | Ghrelin measured 120 minutes post meal consumption
  Ghrelin (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on ghrelin levels (T180) | Ghrelin measured 180 minutes post meal consumption
  Ghrelin (pmol/L)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on appetite (T30) | Visual Analogue Scale for Appetite (VAS-A) collected 30 minutes after meal consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score, the greater the level of appetite)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on appetite (T60) | Visual Analogue Scale for Appetite (VAS-A) collected 60 minutes after meal consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score, the greater the level of appetite)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on appetite (T120) | Visual Analogue Scale for Appetite (VAS-A) collected 120 minutes after meal consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score, the greater the level of appetite)
To assess the acute effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on appetite (T180) | Visual Analogue Scale for Appetite (VAS-A) collected 180 minutes after meal consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score, the greater the level of appetite)

SECONDARY OUTCOMES:
To assess the perception of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake. Subjective analysis including Visual Analogue Scale for Perception and Palatability (VAS-P). | VAS for Perception and Palatability collected immediately after meal consumption
  Scores range from 0 to 100 (the higher the score, the lower the palatability)
To assess the effects of oat porridge, whey protein isolate, potato protein isolate, and meal replacement shake on food intake ad libitum, 3 hours after the intervention meal consumption. | Ad libitum food intake was assessed 3 hours post breakfast intervention meal consumption
  Consecutive meal intake was assessed by measuring the weight in grams and calculating the energy content in Kcal of the food consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Gulrez Zariwala, PhD, Principal Investigator — University of Westminster
Locations (1):
- Centre for Nutraceuticals School of Life Sciences, University of Westminster, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan MAB, Hashim MJ, King JK, Govender RD, Mustafa H, Al Kaabi J. Epidemiology of Type 2 Diabetes - Global Burden of Disease and Forecasted Trends. J Epidemiol Glob Health. 2020 Mar;10(1):107-111. doi: 10.2991/jegh.k.191028.001. PMID 32175717
- [Background] Guo H, Guo Q, Li Z, Wang Z. Association between different GLP-1 receptor agonists and acute pancreatitis: case series and real-world pharmacovigilance analysis. Front Pharmacol. 2024 Nov 13;15:1461398. doi: 10.3389/fphar.2024.1461398. eCollection 2024. PMID 39605914
- [Background] Ismail I, Hwang YH, Joo ST. Meat analog as future food: a review. J Anim Sci Technol. 2020 Mar;62(2):111-120. doi: 10.5187/jast.2020.62.2.111. Epub 2020 Mar 31. PMID 32292920
- [Background] Monami M, Nreu B, Scatena A, Cresci B, Andreozzi F, Sesti G, Mannucci E. Safety issues with glucagon-like peptide-1 receptor agonists (pancreatitis, pancreatic cancer and cholelithiasis): Data from randomized controlled trials. Diabetes Obes Metab. 2017 Sep;19(9):1233-1241. doi: 10.1111/dom.12926. Epub 2017 Jun 20. PMID 28244632
- [Background] Patel S. Emerging trends in nutraceutical applications of whey protein and its derivatives. J Food Sci Technol. 2015 Nov;52(11):6847-58. doi: 10.1007/s13197-015-1894-0. Epub 2015 Jun 9. PMID 26884639
- [Background] Santesso N, Akl EA, Bianchi M, Mente A, Mustafa R, Heels-Ansdell D, Schunemann HJ. Effects of higher- versus lower-protein diets on health outcomes: a systematic review and meta-analysis. Eur J Clin Nutr. 2012 Jul;66(7):780-8. doi: 10.1038/ejcn.2012.37. Epub 2012 Apr 18. PMID 22510792
- [Background] Zushin PH, Wu JC. Evaluating the benefits of the early use of GLP-1 receptor agonists. Lancet. 2025 Jan 18;405(10474):181-183. doi: 10.1016/S0140-6736(24)02255-4. Epub 2024 Nov 12. No abstract available. PMID 39547251
- See also: NHS. (2023). Obesity - Treatment — http://www.nhs.uk/conditions/obesity/treatment/
- See also: WHO. (2024). Obesity and overweight. World Health Organization. — http://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight
- See also: WHO. (2015). World health statistics 2015. World Health Organization — https://www.who.int/docs/default-source/gho-documents/world-health-statistic-reports/world-health-statistics-2015.pdf